CLINICAL TRIAL: NCT04555928
Title: Measuring Pain Intensity in Older Patients: A Comparison of Five Scales
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sasikaan Nimmaanrat, Department of Anesthesiology, Prince of Songkla University
Other Study IDs: REC.63-050-8-1
Record Dates: First submitted 2020-08-28; First posted 2020-09-21 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Pain Measurement; Geriatric Patients
Keywords: pain measurement, geriatric patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is a prospective cohort (survey) study. It has no intervention.

SUMMARY:
Pain intensity is commonly measured in research and clinical settings.1 Different pain intensity domains can be assessed, depending on the specific goals of the researcher or clinician. These include current pain, and recalled average pain, least pain and worst pain in the past 24 hours or 7 days. Although average pain (in the past 24 hours or 7 days) is arguably the most common pain intensity domain assessed by researchers and clinicians, some researches indicate that in chronic pain samples, worst pain is more strongly associated with disability than average pain.2 Thus, while current pain is likely the most appropriate pain intensity domain in acute pain contexts (e.g., during medical procedures), both average and worst pain are important domains to consider assessing the chronic pain context. As such, research to understand the most reliable and valid measures for assessing these domains in different pain populations is critical for both researchers and clinicians.

DETAILED DESCRIPTION:
The majority of clinical guidances, such as those of the American Pain Society (APS) recommend routine pain measurement. Pain intensity can be assessed by using self-report measures, observational measures, and/or physiological measures. Among these, self-report measures are regarded as the gold standard because pain severity is always a subjective experience.3 The Australian and New Zealand Society for Geriatric Medicine has issued a position statement emphasizing that self-report should be the gold standard, while observational and behavioral scales should be employed for individuals unable to reliably report pain due to cognitive or communication deficits.4 Self-reporting requires an individual to communicate this personal unpleasant sensory and emotional experience as well as to process external information.5 The three most commonly used self-report pain intensity measurement tools are the Visual Analog Scale (VAS), Numerical Rating Scale (NRS), and the Verbal Rating Scale (VRS). The Faces Pain Scale-Revised (FPS-R), originally developed for use with children, is increasingly used in pediatric populations as well as populations who might find the complexity of the VAS, NRS, and even the VRS challenging (e.g., individuals with very low educational levels or individuals with cognitive deficits.6 Each of these four scales has its strengths and weaknesses, and there is no single scale recommended for use with all patient groups in all situations.7 As indicated previously, faces pain scales such as the FPS-R were originally developed for use in young children and adults with low educational levels or cognitive deficits. However, concerns have been expressed that faces pain scales may not be as valid as the other measures for assessing pain intensity only, as they may also reflect the patient's emotional response to the pain.8 In addition, there are inconsistencies in the way different individuals interpret measurement tools9; the most suitable tool for any population may depend on that population's age, education level, or culture.10 Although the VAS has traditionally been thought to be sensitive to small changes in pain than the other commonly used pain intensity measures, research suggests that it is more difficult to comprehend than other tools, especially for the elderly and those with cognitive impairments.11 In July 2019, the world population reached 7.7 billion people. The world population is estimated to reach 8 billion people in 2023 and 10 billion people in the year 2056. Thailand is the 20th country among the top 20 largest countries by population.12 As life expectancy increases, the geriatric population is increasing. The number of people older than 60 years of age has tripled since 1950 and exceeded 700 million in 2006. It is estimated that the older population will reach 2.1 billion by the year 2050.13 Thus, we can anticipate in the years and decades ahead, many more elderly patients will be receiving health care.

Given decreases in both physical function and cognitive abilities, geriatric people are considered vulnerable. Although pain is an important issue for this population, inadequate attention has been provided to its assessment and management. Uncontrolled pain can be physically and psychologically harmful. As a result, the quality of life and ability to function in the elderly is at risk because of the inadequate or inappropriate treatment of pain. Importantly, valid and reliable pain assessment is central to the appropriate treatment of pain.14 In order to provide the highest quality of health care, health care providers should be able to recognize, assess and manage pain appropriately.15 A number of studies have been conducted in otherwise healthy and pain older adults to evaluate the psychometric properties of commonly used pain assessment tools as well as preferences for a tool of choice. For example, 167 patients with a mean age of 80.5 years were included in a study to evaluate the utility and validity of 3 different pain rating scales: a VAS, a Graphic Rating Scale (GRS), and a NRS. They found that all 3 pain rating scales were valid for assessing pain intensity in geriatric patients. However, the agreement between verbally expressed experience and the rated experience of pain tended to decrease with advancing age.15 A quasi-experimental study was conducted in a group of younger and older (age 65-94) healthy volunteers. Responses of subjects to induced noxious thermal stimuli were measured with 5 pain scales: a vertical VAS, a 21-point NRS, an 11-point VNS (e.g., participants were instructed to give their responses to a VRS verbally rather than on a paper-and-pencil form), an 11-point Verbal Descriptor Scale (VDS) and a FPS. All 5 scales were found to be reliable and valid across all ages, although the VDS was preferred over the other measures in the older adults, including those with mild to moderate cognitive impairment.16 A study conducted in nursing home residents with varying degrees of cognitive impairment found that the association among five different scales (VRS, NRS, FPS, color analogue scale and mechanical VAS] was strong among participants with no to moderate cognitive impairment, but poor for those severely impaired. The findings also revealed no systematic differences in the means of the pain scores between the measures as a function of cognitive status.11 Cognitively impaired and intact nursing home residents with mean age of 78.4 years participated in a study to compare 4 standard pain intensity instruments (a VRS from the McGill Pain Questionnaire, Wong-Baker Pain Faces Scale, a VAS and a VRS). They concluded that the VRS was the most useful for assessing pain intensity in this sample.17 A study performed in a sample of Chinese postoperative adult patients who presented without and with mild cognitive impairment compared the psychometric properties of 5 pain intensity scales (VDS, NRS, FPS, 21-point Box Scale (BS-21), Colored Analogue Scale [CAS]). The findings supported the validity of all 5 pain scales in the sample, including those with mild cognitive impairment. However, a slight the FPS appeared to evidence somewhat stronger validity, followed by the VDS and NRS.18 A study to compare the VAS, VDS, Pain Thermometer (PT) and NRS in 40 elderly women who experienced chronic arthritic pain. Almost half of the subjects rated the Pain Thermometer as the easiest and most accurate reflection, followed by the VDS, VAS and NRS.19 A preliminary study in younger (21-55 years old) and older (65-87 years old) adults with arthritic pain who were administered different rating scales before and after joint injection demonstrated that Iowa Pain Thermometer (IPT) was the most sensitive to the effects of the injection on pain intensity, had the lowest failure rate, and was the most preferred, when compared to the NRS, verbal NRS (VNS), FPS, and VAS.20 A study in older minority adults demonstrated that samples with intact cognitive function and cognitive impairment were able to use each of the 4 pain scales [IPT, NRS, Verbal Descriptor Scale (VDS) and Faces Pain Scale-Revised (FPS-R)].21 Another study was done in a sample of African American older individuals with both intact and impaired cognitive function. The findings indicated that cognitive impairment did not interfere with the older adults to use any of the tools evaluated (FPS, VDS, NRS, and IPT). However, both the cognitively impaired and intact groups preferred the FPS over the other measures.22 A descriptive correlational designed study was carried out in a sample of cognitively intact and cognitively impaired older adults to determine the reliability and validity of the FPS, VDS, NRS and IPT. The average Mini Mental State Exam (MMSE) score was 16, with a range of 1-29. Eighty-five percent of the sample had some degree of cognitive impairment (e.g., a MMSE score of 24 or lower) while 15% classified as being cognitively intact. Concurrent validity of the VDS, NRS and IPT was supported in the entire sample. However, the FPS demonstrated weak correlations with other scales in the cognitively impaired group. Test-retest reliability at a 2-week interval was acceptable in the cognitively intact group and unacceptable for all in the cognitively impaired group.23 One hundred and seventy-seven subjects aged 65 years or older were asked to rate their pain intensity by using FPS-R and pain thermometer (PT) in 5 hypothetical painful situations (Geriatric Painful Events Inventory) at 2 different times. The results showed that the pain intensity ratings reported with FPS-R and PT were very similar. Also, all of the participants preferred the FPS-R over the PT, regardless of age or gender.24 Five commonly used pain scales (a VAS, a vertical VAS, an 11-point BS, and a VDS) were studied in younger and older patients with chronic pain. It was found that Box-21 was an excellent choice across different age groups, although patients older than 75 years preferred the verbal descriptor scale.10 Comparing the 11 face modified version of the McGrath nine face Faces Pain Scale (FPS) with an 11-point NRS in sample of Korean older adults 85 years old or more, Kim and colleagues found that the 11-point NRS was appropriate in this population.25 Difficulties with the VAS among surgical elderly patients were identified including high rates of unscorable data and low face validity. The authors concluded that its use in elderly postoperative patients should be discouraged.26 Overall, this body of research indicates that all of the most commonly used measures of pain intensity, including the VAS, VRS, NRS, and faces scales (the FPS and FPS-R are the faces scales examined most often) tend to be valid for measuring pain intensity in cognitively intact elderly healthy and patient populations, although when problems do emerge, the VAS is the scale found to have more problems (including higher failure rates) than the other scales. In elderly individuals with cognitive deficits, fewer problems tend to emerge as the scales become more simple, with the most valid and useful scales being, in order, the FPS/FPS-R, the VRS, the 0-10 NRS, and the VAS. Moreover, the simpler scales tend to be preferred over the more complicated scales.

However, whether these findings replicate in a sample of elderly patients experiencing pain in Thailand is not known; to our knowledge, no research has yet compared the psychometric properties of the most commonly used pain intensity scales in a sample of elderly individuals from Thailand. As a result, it is not possible to make recommendations regarding which scales to use when performing research or providing health care in elderly Thai patients, including those who are do and do not have cognitive deficits and have more or less education.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old.
* Endorsing having at least some pain in the past week, from any diagnosis.
* Can speak and write in Thai, as determined by an ability to answer details about demographic information
* No motor deficits in the hands that would interfere with their ability to respond to a paper-and-pencil questionnaire

Exclusion Criteria:

* Lack of fluency in Thai
* Neurological disorder or psychiatric illness that would interfere with participation or ability to provide informed consent
* Refusal to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This quantitative-descriptive cross sectional study will be performed in Songklanagarind Hospital, Thailand, recruiting patients with pain from different inpatient wards and outpatient clinics, including the (1) pain clinic, (2) orthopedic clinic, (3) orthopedic wards, (4) rehabilitation clinic, (5) radiotherapy clinic, (6) oncology clinic, (7) internal medicine wards, (8) surgical wards, (9) trauma ward, (10) gynecological ward and (11) private wards.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Psychometric properties (validity, reliability, and utility) of Verbal Numerical Rating Scale (VNRS) 0-10 | September 2020 until August 2021
  Verbal Numerical Rating Scale or VNRS consists of 0-10 when 0 represents no pain and 10 represents worst pain imaginable. Patients are asked to rate his/her pain verbally.
Psychometric properties (validity, reliability, and utility) of Visual Analog Scale (VAS) 0-10 | September 2020 until August 2021
  Visual Analog Scale or VAS is a 10-cm line where the end of the left side represents no pain and the end of the right side represents worst pain imaginable. The VAS line has no number at all. Patients are asked to draw a mark on the line where it represents their pain.
Psychometric properties (validity, reliability, and utility) of Numerical Rating Scale (NRS) 0-10 | September 2020 until August 2021
  Numerical Rating Scale or NRS is a 10-cm line with numbers 0-10 on it. Zero is on the end of the left side representing no pain while 10 is on the end of the right side representing worst pain imaginable. Each centimeter of the line has a number. Patients are asked to mark on the line.
Psychometric properties (validity, reliability, and utility) of Faces Pain Scale (FPS) 6 faces | September 2020 until August 2021
  Faces Pain Scale or FPS consists of 6 faces. Pain severity increases from the left to the right. Patients are asked to mark on the face representing their pain.
Psychometric properties (validity, reliability, and utility) of Verbal Rating Scale (VRS) 6 words | September 2020 until August 2021
  Verbal Rating Scale or VRS consists of 6 descriptors from left to right: no pain, very mild pain, mild pain, moderate pain, severe pain, very severe pain.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962